CLINICAL TRIAL: NCT06120452
Title: A Clinical Trial to Evaluate the Effectiveness of an Acne Serum in Improving Facial Acne and Post-Acne Pigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rael (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20355
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test arm: Acne Serum (Experimental): Participants will use the serum after cleansing and toning every morning for 8 weeks (56 days).
  Interventions: Other: Rael Miracle Clear Complete Acne Serum

INTERVENTIONS:
Other: Rael Miracle Clear Complete Acne Serum — This acne serum contains the following ingredients:
  1.5% Salicylic acid. 2% Niacinamide. 0.5% Zinc Pyrrolidone Carboxylic Acid (PCA). Hyaluronic Acid.

SUMMARY:
This study will evaluate the efficacy of the Rael Miracle Clear Complete Acne Serum product in improving facial acne and post-acne pigmentation. This study will last for 56 days. The study will be conducted as a single-arm trial where all participants will use the test products. Participants will be required to complete questionnaires at Baseline, Day 1, Day 3, Day 7, Day 14, Day 28, and Day 56. Photos will be taken at Baseline, Day 28, and Day 56. The photos from Baseline and Day 56 will undergo expert skin grading

ELIGIBILITY:
Inclusion Criteria:

* Female. Age 18+. Currently experiencing mild to moderate acne issues. Generally healthy -and not living with any uncontrolled chronic disease.

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.

Anyone currently using an oral and/or topical prescription acne treatment. Anyone unwilling to stop using their current acne supplements. Anyone with known severe allergic reactions. Anyone unwilling to avoid excessive sun exposure. Anyone who is breastfeeding, pregnant, or attempting to become pregnant. Anyone unwilling to follow the study protocol. Anyone who identifies as having sensitive skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in the appearance of facial acne. [Timeframe: Baseline to Day 56] | 56 days
  Before and after photos will undergo virtual skin grading by a board-certified dermatologist to assess this change.
  Participants will also complete questionnaires rating the appearance of their facial acne. Questionnaires will use a 5-point Likert scale, with 0 indicating the less favourable response and 5 indicating the most favourable response.
Changes in the appearance of post-acne pigmentation. [Timeframe: Baseline to Day 56] | 56 days
  Before and after photos will undergo virtual skin grading by a board-certified dermatologist to assess this change.
  Participants will also complete questionnaires rating the appearance of their post-acne pigmentation. Questionnaires will use a 5-point Likert scale, with 0 indicating the less favourable response and 5 indicating the most favourable response.

SECONDARY OUTCOMES:
Changes in facial skin hydration. [Timeframe: Baseline to Day 56] | 56 days
  Before and after photos will undergo virtual skin grading by a board-certified dermatologist to assess this change.
  Participants will also complete questionnaires rating their perception of facial skin hydration. Questionnaires will use a 5-point Likert scale, with 0 indicating the less favourable response and 5 indicating the most favourable response.
Changes in facial skin softness. [Timeframe: Baseline to Day 56] | 56 days
  Participants will complete questionnaires rating their perception of facial skin softness. Questionnaires will use a 5-point Likert scale, with 0 indicating the less favourable response and 5 indicating the most favourable response.
Changes in facial skin texture. [Timeframe: Baseline to Day 56] | 56 days
  Before and after photos will undergo virtual skin grading by a board-certified dermatologist to assess this change.
  Participants will also complete questionnaires rating their perception of facial skin texture. Questionnaires will use a 5-point Likert scale, with 0 indicating the less favourable response and 5 indicating the most favourable response.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided